CLINICAL TRIAL: NCT02953899
Title: Piloting the Addition of Contingency Management to Best Practice Counselling as an Adjunct Treatment for Rural and Remote Disordered Gamblers
Brief Title: Contingency Management as an Adjunct Treatment for Rural and Remote Disordered Gamblers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lethbridge (Other)
Collaborators: Rural Development Network (Unknown)
Responsible Party: Principal Investigator, Darren R. Christensen, Chair in Gambling, Assistant Professor, University of Lethbridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-080
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Gambling Disorder
Keywords: Internet; Contingency Management; Gambling Disorder; Rural
MeSH Terms: conditions — Gambling | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contingency Management (Experimental): This is a treatment where participants earn points for treatment attendance and for providing evidence of gambling abstinence. These points are added to study accounts that can be redeemed for goods and services available at a variety of on-line businesses (e.g., Amazon, Walmart, etc.). Submission of evidence of gambling behaviour or non-attendance at an on-line counselling session re-sets subsequent points to the starting level. The CM procedure is implemented as part of the CBT counselling session.
  Interventions: Behavioral: Contingency Management
- Cognitive Behavioural Therapy (Active Comparator): CBT is currently considered "best practice" for the treatment of problem gambling, as noted in the National Health and Medical Research Council (Australia) endorsed Clinical Guidelines for problem and pathological gambling treatment (Problem Gambling Research and Treatment Centre, 2011). CBT is typically a semi-structured approach for delivering cognitive behavioural therapy addressing the participant's experiences, thoughts, and emotions relating to their gambling and substance use. Techniques include psychoeducation, behavioural interventions, and cognitive strategies. Participants are expected to attend on-line counselling sessions three times a week for approximately 12 weeks. All participants will receive individual counselling from an experienced counsellor/therapist.
  Interventions: Behavioral: Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Contingency Management — In addition to Cognitive Behavioural Therapy, this intervention uses small incentives to reinforce study attendance and gambling abstinence.
  Arms: Contingency Management
Behavioral: Cognitive Behavioural Therapy — This intervention uses psychoeducation, behavioural strategies, and cognitive restructuring to assist the participant in their efforts to become abstinent from gambling.
  Arms: Cognitive Behavioural Therapy

SUMMARY:
The purpose of this project is to pilot contingency management as an adjunct treatment to counselling as usual using internet delivered video-conferencing applications for remote disordered gamblers. This project further investigates the impact of adding contingency management to counselling to improve counselling attendance and retention and uses internet-delivered approaches to assist rural and remote disordered gamblers gain access to counselling treatments.

DETAILED DESCRIPTION:
The chosen methodology is a randomised clinical trial where participants are allocated into one of two conditions; Contingency Management and Cognitive Behavioural Therapy (CM+), or Cognitive Behavioural Therapy alone (CBT) for the treatment of disordered gambling. Participants will experience a battery of tests pre- and post-treatment examining clinical, psychological, and behavioural issues, including co-morbid substance use. Alberta Rural Development Network (ARDN) affiliates will be provided with information regarding how participants can access the Qualtrics study site (e.g., an on-line survey hosting company) and will be individually directed to the study site by the principal investigator to complete the consent form and the base-line assessments. Counselling will be provided free of charge using Skype or Facetime video-conferencing internet applications. Participation in each condition will last 14 weeks: 12 weeks for treatment, and 2 weeks of assessments (one week prior to treatment and one week post treatment). Pre-treatment assessments (including demographic information) will take approximately 30-45 minutes, as will the post-treatment assessments. The progress check-ups by the Principal Investigator will take 5 to 10 minutes. A subset of treatment seekers, counsellors, and community/project stakeholders (e.g., ARDN affiliates) will also be chosen to participate in qualitative interviews to explore their experiences as well as their perceptions regarding the utility of the program for residents of rural and remote areas. The qualitative interviews will take approximately 30-60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* capable of providing written consent,
* received a diagnosis of gambling disorder (American Psychiatric Association, 2013),
* gambled within the last month,
* live in a rural or remote location, and
* speak English

Exclusion Criteria:

* Medically unmanaged psychiatric or neurological disorder(s) except for disordered gambling

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Gambling Abstinence | 12 weeks
  The total number of sessions that a participant provided evidence of gambling abstinence in the study

SECONDARY OUTCOMES:
Session Attendance | 12-weeks
  The total number of sessions that a participant attended the study
Study Retention | 12-weeks
  The total number of weeks that a participant attended the study

CONTACTS AND LOCATIONS:
Overall Officials: Darren R Christensen, PhD, Principal Investigator — University of Lethbridge
Locations (1):
- University of Lethbridge, Lethbridge, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Only the research team will have access to the individual participant data

REFERENCES:
- [Derived] Christensen DR, Witcher CSG, Leighton T, Hudson-Breen R, Ofori-Dei S. Piloting the addition of contingency management to best practice counselling as an adjunct treatment for rural and remote disordered gamblers: study protocol. BMJ Open. 2018 Apr 3;8(4):e018804. doi: 10.1136/bmjopen-2017-018804. PMID 29615445